CLINICAL TRIAL: NCT06053164
Title: Ambulatory Oxygen Therapy for Individuals With Mild-to-moderate Interstitial Lung Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Boehringer Ingelheim Collaboration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00128503
Record Dates: First submitted 2023-08-03; First posted 2023-09-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Fibrotic Interstitial Lung Disease
Keywords: Exertional Oxygen; Ambulatory Oxygen; Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Educational Status; Palliative Care

STUDY DESIGN:
Intervention Model Description: Single-blind open-label randomized control
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind investigation, investigator and assessors will be blinded to the condition/treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Usual Care (No Intervention): 8 weeks of usual care with no supplemental oxygen provided
- Arm 2 - Exertional Oxygen (Experimental): 8 weeks of portable oxygen use (from a concentrator) during exertion
  Interventions: Drug: Exertional Oxygen
- Arm 3 - Exertional Oxygen + Support (Experimental): 8 weeks of portable oxygen use (from a concentrator) during exertion, plus additional phone calls with a respiratory educator and educational material
  Interventions: Drug: Exertional Oxygen; Behavioral: Education and Support

INTERVENTIONS:
Drug: Exertional Oxygen — Use of a portable oxygen concentrator for exertional activities lasting >2 minutes
  Other Names: Supplemental oxygen, ambulatory oxygen
  Arms: Arm 2 - Exertional Oxygen; Arm 3 - Exertional Oxygen + Support
Behavioral: Education and Support — Participants will receive disease-specific educational material (Living Well with Pulmonary Fibrosis: Oxygen), and will have scheduled phone appointments with a certified respiratory educator after 1, 3, and 5 weeks of oxygen therapy in order to address individual barriers to oxygen use and facilitate the optimal use of portable oxygen.
  Arms: Arm 3 - Exertional Oxygen + Support

SUMMARY:
The investigators plan to conduct a study to find out if giving portable oxygen therapy (during physical activity) to patients with interstitial lung disease will improve quality of life, exercise tolerance, shortness of breath, and blood vessel function. Oxygen will be provided for a period of 8 weeks. Additionally, the investigators plan to investigate if it is helpful to deliver individualized support when providing oxygen therapy, through check-in phone calls with a respiratory therapist and by providing additional educational material.

DETAILED DESCRIPTION:
Brief Summary:

The investigators plan to conduct a study to find out if giving portable oxygen therapy (during physical activity) to patients with interstitial lung disease will improve quality of life, exercise tolerance, shortness of breath, and blood vessel function. Oxygen will be provided for a period of 8 weeks. Additionally, the investigators plan to investigate if it is helpful to deliver individualized support when providing oxygen therapy, through check-in phone calls with a respiratory therapist and by providing additional educational material.

Detailed Description:

BACKGROUND

Interstitial lung disease (ILD) is comprised of a group of pulmonary diseases that are characterized by inflammation and/or lung parenchymal fibrosis. Individuals with ILD may be normoxic at rest; however, underlying impairments in gas exchange can contribute to a reduction in oxygen saturation (SpO2) during exertion. Hypoxemia can cause inflammation and cardiovascular dysfunction, which could lead to cardiac events. A recent study found that 78% of ILD patients had cardiovascular comorbidity, which was predictive of death within this ILD cohort.

Oxygen therapy is used in patients with advanced lung disease with resting hypoxemia; however, there is limited evidence regarding its clinical efficacy. Furthermore, there is little support to describe the benefit of ambulatory oxygen therapy in individuals with lung disease who are normoxemic at rest but become hypoxemic with exertion. Accordingly, thresholds for the prescription of oxygen therapy vary between (and within) health districts and geographical regions, and individuals who might benefit from supplemental oxygen typically do not qualify for funding of oxygen therapy under unclear guidelines. Furthermore, data from studies in patients with chronic obstructive pulmonary disease (COPD) are often extrapolated for use in guiding oxygen therapy in patients with ILD, which is likely inappropriate considering recent research demonstrated that individuals with fibrotic ILD experience greater hypoxemia than those with COPD during the 6-minute walk test (6MWT).

Oxygen therapy may be beneficial in reducing inflammation, oxidative stress, and pulmonary artery pressure, all of which are elevated in ILD. Furthermore, a reduction in dyspnea during exercise with exertional oxygen therapy might increase daily physical activity, exercise tolerance, and reduce overall sedentary time, which would have a positive effect on vascular function. These postulated outcomes, however, are confounded by various practical, psychological, and social challenges associated with use of an oxygen concentrator, as well as challenges with proper titration of oxygen levels (accurately targeting appropriate SpO2) in relation to exertional intensity. Paradoxically, if the flow of oxygen is too high, activation of inflammatory and oxidative pathways may inhibit the benefits related to the alleviation of hypoxemia. Thus, integration of patient-specific disease support tools is essential when initiating oxygen therapy to ensure appropriate oxygenation during exertion.

OBJECTIVE To assess the feasibility of oxygen therapy, education, and support for individuals with fibrotic interstitial lung disease and exertional hypoxemia. As a secondary objective, the effects of exertional oxygen therapy and support on physical activity, vascular function, and health-related quality of life in individuals with fibrotic interstitial lung disease will be investigated.

PRIMARY AND SECONDARY ENDPOINTS

Health related quality of life as assessed by the EQ-5D-5L and the K-BILD Exercise tolerance, assessed by 6MWD while breathing room air Daily physical activity and sedentary time as assessed by a remote monitor. Dyspnea, as measured by the Dyspnea 12 questionnaire Cough using the visual analog scale (VAS) and cough score (measured by Leicester Cough Questionnaire; LCQ) Vascular function, measured by flow mediated dilation (FMD) of the brachial artery Pulmonary artery systolic pressure (PASP) measured by cardiac echocardiography Cardiac systolic and diastolic function assessed by cardiac echocardiography Systemic inflammation

STUDY DESIGN

Single-blind (assessment team) open-label randomized control

TRIAL TREATMENT

Participants will be randomized into one of three arms:

Control:

(Arm 1) 8 Weeks of usual care (n=20)

Treatment:

(Arm 2) 8 Weeks of supplemental oxygen(n=20)

(Arm 3) 8 Weeks of supplemental oxygen plus educational materials and scheduled support (n=20)

All: 2-week baseline prior to intervention and 2-week washout post-intervention to document carry-over effect of intervention.

DURATION

Seven sessions will be completed over a 13-week period.

TIMELINE

Visit 1) Participant enrollment, medical history, standard pulmonary function test (PFT) and 6-minute walk test (6MWT); followed by 1-week for collection of baseline physical activity and SpO2. During this visit, participants will be provided a wrist-worn activity monitor and a finger-worn pulse oximeter. This visit will take approximately 3 hours.

Visit 2) Doppler measurements of systemic vascular function (flow mediated dilation) will be measured at rest while breathing room air. A small sample of venous blood will be taken to analyze inflammatory levels and reactive oxygen species. Participants will fill out questionnaires relating to health-related quality of life, dyspnea, and cough. Finally, participants will perform tests of lung diffusing capacity for carbon monoxide (DLCO) under three different conditions: seated, supine, and during exercise at 40W on a cycle ergometer.

Visit 3) One to three days after Visit 2, participants will return for the second day of pre-intervention baseline testing. An echocardiographic exam will be completed to determine pulmonary artery systolic pressure as well as systolic and diastolic function in the left and right ventricles of the heart. To enhance the Doppler signal during the cardiac ultrasound, agitated saline contrast will be used. Two 6-minute walk tests will then be completed, separated by half an hour. This visit will take approximately 2 hours. Following this day, participants will be randomized into one of three arms for an 8-week intervention.

Eight-week intervention, randomized into one of:

* No oxygen
* Exertional oxygen
* Exertional oxygen + additional support

Visit 4) Repeat Day 2 protocol. Visit 5) Repeat Day 3 protocol.

Two-week washout period

Visit 6) Repeat Day 2 protocol. Visit 7) Repeat Day 3 protocol.

The total duration of time spent for each participant will be approximately 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with fibrotic ILD (all sub-groups of ILD) who have normal oxygen saturation at rest (SpO2 > 90%) but develop exertional hypoxemia as demonstrated by a SpO2 = 80-89% with activity (measured during 6MWT).

Exclusion Criteria:

* Use of home oxygen therapy within the previous year for the management of ILD, co-morbid conditions that may require oxygen therapy (such as COPD, cardiovascular disease, or other illnesses), or individuals that require the use of non-invasive ventilation. Additionally, individuals with significant cardiovascular, metabolic, neuromuscular or any other disease that could contribute to dyspnea or abnormal cardiopulmonary responses to exercise will be excluded. Individuals with musculoskeletal injuries that prevent them from completing cycle ergometry exercise trials and ambulation will also be excluded. Individuals with peripheral vascular disease will be excluded from measurement of vascular function (flow mediated dilation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of investigation | 2 years
  Number of patients recruited and completing the protocol in each arm
Exercise tolerance | Before and immediately after the intervention
  6 minute walk distance
Health Related Quality of Life, (EuroQol-5 Dimension-5 Level; EQ-5D-5L) | Before and immediately after the intervention
  Questionnaire for Health-Related Quality of Life. Possible Range = 5-25; 5 = 11111 (no problems on any dimension); 25 = 55555 (extreme problems on all dimensions)
Health Related Quality of Life, (King's Brief Interstitial Lung Disease Questionnaire; KBILD) | Before and immediately after the intervention
  Health status questionnaire. Domain and total score ranges are 0-100; 100 represents best health status

SECONDARY OUTCOMES:
Dyspnea (Dyspnea-12 Questionnaire) | Before and immediately after the intervention
  Range from 0-36, 0 represents no breathlessness and 36 represents maximal severity
Vascular function | Before and immediately after the intervention
  Flow-mediated dilation
Cough (Leicester cough questionnaire; LCQ) | Before and immediately after the intervention
  Quality of life measure of chronic cough. Range from 3-21, lower score indicating greater impairment of health status due to chronic cough
Pulmonary Artery Pressure | Before and immediately after the intervention
  Echocardiography-derived pulmonary artery systolic pressure
Cardiac Output | Before and immediately after the intervention
  Assessed by echocardiography (L/min)
Systemic Inflammation | Before and immediately after the intervention
  C-Reactive Protein (CRP, venous blood, mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Stickland, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khor YH, Holland AE, Goh NSL, Miller BR, Vlahos R, Bozinovski S, Lahham A, Glaspole I, McDonald CF. Ambulatory Oxygen in Fibrotic Interstitial Lung Disease: A Pilot, Randomized, Triple-Blinded, Sham-Controlled Trial. Chest. 2020 Jul;158(1):234-244. doi: 10.1016/j.chest.2020.01.049. Epub 2020 Feb 28. PMID 32113924
- [Background] Johannson KA, Pendharkar SR, Mathison K, Fell CD, Guenette JA, Kalluri M, Kolb M, Ryerson CJ. Supplemental Oxygen in Interstitial Lung Disease: An Art in Need of Science. Ann Am Thorac Soc. 2017 Sep;14(9):1373-1377. doi: 10.1513/AnnalsATS.201702-137OI. PMID 28644693
- [Background] Visca D, Mori L, Tsipouri V, Fleming S, Firouzi A, Bonini M, Pavitt MJ, Alfieri V, Canu S, Bonifazi M, Boccabella C, De Lauretis A, Stock CJW, Saunders P, Montgomery A, Hogben C, Stockford A, Pittet M, Brown J, Chua F, George PM, Molyneaux PL, Margaritopoulos GA, Kokosi M, Kouranos V, Russell AM, Birring SS, Chetta A, Maher TM, Cullinan P, Hopkinson NS, Banya W, Whitty JA, Adamali H, Spencer LG, Farquhar M, Sestini P, Wells AU, Renzoni EA. Effect of ambulatory oxygen on quality of life for patients with fibrotic lung disease (AmbOx): a prospective, open-label, mixed-method, crossover randomised controlled trial. Lancet Respir Med. 2018 Oct;6(10):759-770. doi: 10.1016/S2213-2600(18)30289-3. Epub 2018 Aug 28. PMID 30170904